CLINICAL TRIAL: NCT04593225
Title: Effectiveness of Virtual Multicomponent Treatment for Chronic Fatigue Syndrome: VIRTUAL SFCAMINA STUDY
Brief Title: Effectiveness of VIRTUAL SFCAMINA STUDY
Acronym: SFCAMINA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)490/2020
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Chronic Fatigue Syndrome
Keywords: multicomponent treatment; Chronic Fatigue Syndrome; pain neuroscience education; therapeutic exercise; cognitive behavioural therapy; mindfulness; randomized controlled trial
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Single-blind, parallel-group, randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU + multicomponent treatment VIRTUAL SFCAMINA (Experimental): VIRTUAL SFCAMINA is a multicomponent non-pharmacological program based on Pain Neuroscience Education (PNE), therapeutic exercise, Cognitive Behavioural Therapy (CBT) and Mindfulness Training
  Interventions: Behavioral: TAU + multicomponent treatment VIRTUAL SFCAMINA
- Treatment as Usual (TAU) (Active Comparator): Treatment-as-Usual (TAU) consisted of the prescribed drugs adapted to the symptomatic profile of each patient and basic face to face and written advice on PNE and aerobic exercise adapted to the physical capacities of the patients at the beginning of the study.patient
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: TAU + multicomponent treatment VIRTUAL SFCAMINA — Group treatment protocol of 12 weekly 60 minute virtual sessions. All sessions include the following ingredients (approx. in the same order): - Pain neuroscience education (15 min.) - Cognitive restructuring (15 min.) - Mindfulness techniques (15 min.) - Physical exercise(15 min.) - Treatment as Usual (TAU) Standard pharmacological treatment usually provided to patients with SFC.
  Arms: TAU + multicomponent treatment VIRTUAL SFCAMINA
Behavioral: Treatment as Usual (TAU) — Treatment-as-Usual (TAU) consisted of the prescribed drugs adapted to the symptomatic profile of each patient and basic face to face and written advice on PNE and aerobic exercise adapted to the physical capacities of the patients at the beginning of the study.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The main objective of this study is to analyse the effectiveness of the VIRTUAL SFCAMINA multicomponent treatment program as coadjuvant of treatmentas- usual (TAU) compared to TAU alone. In this Randomized Controlled Trial (RCT), in addition to evaluating the clinical effects of VIRTUAL SFCAMINA treatment in the short- and long term.

DETAILED DESCRIPTION:
This is a tree-arm RCT focused on the safety and potential effectiveness of the multicomponent program VIRTUAL SFCAMINA as coadjuvant of treatmentas- usual (TAU) vs. TAU alone.

* VIRTUAL SFCAMINA combines multicomponent approach based on Pain Neuroscience Education (PNE), therapeutic exercise, Cognitive Behavioural Therapy (CBT) and Mindfulness training.
* The main hypothesis is that improvement on fatigue of patients with fibromyalgia can be achieved by the direct intervention on mechanisms such as kinesiophobia, fear avoidance and by individualized therapeutic exercise.

ELIGIBILITY:
Inclusion Criteria:

* Meet the Fukuda and Holmes classification criteria for Fatigue Syndrome Chronicle
* Age equal to or greater than 18 years
* Understand and agree to participate in the study
* Sign the informed consent

Exclusion Criteria:

* Terminal clinical conditions or scheduled treatments that may interrupt the study follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2021-12-21 (Estimated); Study Completion 2022-01-21 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Fatigue Inventory (MFI) | Through study completion, an average of 3 months
  Multidimensional Fatigue Inventory (MFI), a 20-item instrument consisting of several subscales including general fatigue and reduced activity. Severe fatigue it is defined as a score of greater than or equal to 13 on the MFI general fatigue subscale or greater than or equal to 10 on the MFI reduced activity subscale. The mean MFI general fatigue scores ranged from 18.3 to 18.8

SECONDARY OUTCOMES:
Tampa Scale for Kinesiophobia (TSK-11) | Through study completion, an average of 3 months
  TSK-11 is used to assess fear of pain and movement. It consists of 11 items, which are answered on a Likert scale of 4 points. Total scores of each scale range from 11 to 44, where higher scores indicate a greater fear of pain and movement.
Hospital Anxiety and Depression Scale (HADS) | Through study completion, an average of 3 months
  HADS is used to quantify the severity of anxiety and depression symptoms. It consists of two dimensions (anxiety and depression) of 7 items each responding on a Likert scale of 4 points. Total scores of each scale (HADS-A and HADSD) range from 0 to 21, where higher scores indicate greater severity of symptoms.
Physical Function of the 36-Item Short Form Survey (SF-36) | Through study completion, an average of 3 months
  Physical Function of the 36-Item Short Form Survey (SF-36) was used to measure physical function.This dimension comprises a total of 10 items, which are answered on a Likert scale of 3 points. Total scores on each scale are then transformed and can range from 0 to 100, with higher scores indicate better physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Mayte Serrat, MSc, Principal Investigator — Vall d'Hebrón Hospital
Locations (1):
- Vall d'Hebrón Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serrat M, Navarrete J, Ferres S, Auer W, Sanmartin-Sentanes R, Nieto R, Neblett R, Borras X, Luciano JV, Feliu-Soler A. Effectiveness of an online multicomponent program (FATIGUEWALK) for chronic fatigue syndrome: A randomized controlled trial. Health Psychol. 2024 Apr;43(4):310-322. doi: 10.1037/hea0001346. Epub 2023 Dec 21. PMID 38127508